CLINICAL TRIAL: NCT04231006
Title: Salvage High Dose Rate Brachytherapy for Local Recurrence in Prostate Cancer: A Phase II Trial
Brief Title: Salvage HDR for Locally Recurrent Prostate Cancer
Acronym: PROSALBRA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Simon Buus, Principal investigator, Aarhus University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1-10-72-218-19
Record Dates: First submitted 2020-01-07; First posted 2020-01-18 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Single arm
  Interventions: Radiation: High dose rate brachytherapy

INTERVENTIONS:
Radiation: High dose rate brachytherapy — High dose rate brachytherapy will be delivered to the site of recurrence within the prostate gland based on MRI and PSMA PET/CT

SUMMARY:
The study offers focal salvage brachytherapy for prostate cancer patients with a local recurrence after primary defintive radiotherapy

DETAILED DESCRIPTION:
The aim of this study is to examine the efficacy and toxicity of focal salvage high dose rate brachytherapy (HDR BT) for patients with locally recurrent prostate cancer after definitive external beam radiotherapy. Furthermore, the investigators want to assess, whether it is feasible to perform salvage HDR BT as a focal treatment based on multiparametric (mp) pelvine MRI and PSMA PET/CT.

ELIGIBILITY:
Inclusion Criteria:

* Man ≥ 18 years, who had definitive EBRT or BT for prostate cancer T1-3b, N0-1, M0
* ≥ 2 years since the end of primary radiotherapy
* PSA recurrence Phoenix criteria (nadir + 2)
* No evidence of regional lymph nodes or distant metastases on PSMA PET/CT
* MRI guided biopsy-proven local recurrence of adenocarcinoma in the prostate gland or seminal vesicles
* GTV identifiable on mpMRI
* No current endocrine therapy
* Plasma testosterone ≥1.75 nm/l
* PSA doubling time ≥ 6 months and ≤ 24 months
* Performance status 0-1
* DAN PSS score ≤ 20
* Maximal urinary flow ≥ 10 ml/s
* Life expectancy > 5 years
* PSA ≤ 10 ug/L at recurrence

Exclusion Criteria:

* Pubic arc interference or major calcifications within the prostate gland.
* Contraindication for spinal or general anaesthesia.
* Conditions indicating that the patient cannot go through the radiation therapy or follow-up, or a condition where the treating oncologist thinks the patient should not participate in the trial, for example due to language problems.
* Inflammatory bowel disease
* Contraindications to 3T MRI
* eGFR < 30 ml/min
* ≥ Gr 3 urinary toxicity at baseline as assessed by CTCAE 4

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2035-03-01 (Estimated)

PRIMARY OUTCOMES:
Time to castration-resistant prostate cancer | 10 years
  The time from intervention until the prostate cancer becomes castration resistant

SECONDARY OUTCOMES:
Erectile dysfunction | 5 years
  Erectile dysfunction as reported by patients in CTCAE PRO
Urinary symptoms | 5 years
  Urinary symptoms as reported by patients in CTCAE PRO
Bowel symptoms | 5 years
  Bowel symptoms as reported by patients in CTCAE PRO

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oncology, Aarhus, Region Midt, Denmark

IPD SHARING:
Plan to Share IPD: No